CLINICAL TRIAL: NCT04834154
Title: Addressing Mental Health Disparities in Spanish Speaking Latina Breast Cancer Patients
Brief Title: Mental Health Disparities in Spanish Speaking Latina Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-57111; NCI-2021-06706 (Other: Clinical Trials Reporting Program (CTRP)); BRS0123 (Other: Stanford OnCore Number)
Record Dates: First submitted 2021-03-22; First posted 2021-04-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Depression, Anxiety; Mindfulness; Sleep Disturbance
Keywords: behavioral intervention; Spanish speaking; Latina; Breast Cancer; Mindfulness
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders; Parasomnias | interventions — Mindfulness; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group visit (Active Comparator): Participants will attend 6 weekly educational and mindfulness sessions
  Interventions: Behavioral: Mindfulness
- Wait list control (Placebo Comparator): Participants will be placed on a wait list
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Mindfulness — 6 weekly 2.0 hour video-conferenced group sessions with the following components: 1) short grounding meditation, 2) check in/review of prior weeks practice and symptoms, 3) educational topic, 3) main meditation, 4) reflection on meditation, and 5) action plan formation
  Other Names: Educational video
  Arms: Mindfulness group visit
Behavioral: Control group — Wait list control
  Arms: Wait list control

SUMMARY:
The purpose of the study is to:Translate a mindfulness program into Spanish for Latina patients with breast cancer.Train a community health worker to facilitate the mindfulness program. Determine if this program is culturally acceptable and feasible, and Obtain pilot data on the program's effectiveness in reducing anxiety and depression

DETAILED DESCRIPTION:
Primary aims of this study are to: 1) translate a behavioral health intervention into Spanish, 2) deliver it to a population of Spanish speaking Latina breast cancer patients, and 3) determine acceptability and feasibility. Secondary aims are to gather preliminary data on anxiety, depression and sleep quality pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self reported diagnosis of invasive breast cancer who has currently or within last 12 months been in active treatment (surgery, chemotherapy, or radiation) or on endocrine therapy
* Self-identified anxiety (persistent worry or nervousness), depression (feeling sad, little interest or pleasure in doing things or hopeless), or sleep disturbance.
* Breast cancer related treatment (surgery, radiation, chemotherapy) or endocrine therapy within the last 12 months
* Self identifies as Spanish speaking
* Self identifies as Latinx / Latina / Latino
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Non-Spanish speaking
* other diagnosis besides invasive breast cancer (ie Ductal carcinoma in situ (DCIS), fibroadenoma, abnormal mammogram but not yet with final diagnosis, non-breast cancer patients)
* comorbid bipolar affective disorder or psychotic disorder (as self-identified by patient after asking "do you have any other psychiatric conditions")
* inability to physically or psychologically attend group sessions, and by discretion of the study coordinator.
* Patients currently participation in stress reduction or mindfulness groups/interventions will be excluded from participation
* Cancer "survivors" if not in active or endocrine treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Acceptability change across session | End of each week for 6 weeks
  The Acceptability scale was developed for this study and is a 5 point Likert scored scale that will be administered after end of each weeks for 6 weeks. There are two questions with scores ranging from "strongly disagree" (score 0), "disagree" (score 1), "neutral" (score 2), "agree" (score 3), and "strongly agree" (score 4). Scores range from 0 to 8 with the higher scores representing greater levels of acceptability. It has 2 additional open ended questions: "What changes did you make in your daily routine as a result of this intervention, if none, why" and "Were there any barriers to making changes you listed on your action plan, if so what were they? The scale takes approximately 5 minutes to complete. Acceptability change will be measured after each session (week 1-6). The mean score with standard deviation for each 6 sessions and acceptability will be reported.
Difference in Feasibility | Through study completion, an average of 1 year
  The Feasibility and Satisfaction scale was developed for this study and is a 5 point Likert scored scale that will be administered at at time of completion of intervention or at time of withdraw (if participant withdraws prior to completion of intervention.) Five questions are scored from "strongly disagree" (score 0), "disagree" (score 1), "neutral" (score 2), "agree" (score 3), and "strongly agree" (score 4). Scores range from 0 to 20 with higher scores representing greater levels of feasibility. Differences in Feasibility will be evaluated and reported. There is also 1 open-ended question "What is the optimal number of visits" with continuous numeric score (participants able to write in number of preferred visits) with higher score representing desire for greater number of visits. The scale takes approximately 5-10 minutes to complete

SECONDARY OUTCOMES:
Differences in Generalized Anxiety Disorder-7 (GAD7) between time points. | Three time points (week 1 and 6 of intervention, and 3 months post intervention.)
  The GAD7 is a well validated seven-item self-administered questionnaire used to measure anxiety. It has 7 questions with Likert scores ranging from "not at all" (score 0), "several days" (score 1), "more than half the days" (score 2), and "nearly every day (score 3).Scores range from 0 to 21 with higher scores indicating higher levels of anxiety, and a cutoff of or above 10 representing high likelihood of generalized anxiety disorder. Difference in GAD-7 measured at three time points (week 1 and 6 of the intervention and 3 months post intervention) will be compared and reported. The scale takes approximately 5-10 minutes to complete
Differences in Center for Epidemiological Studies-Depression (CES-D) between time points. | Three time points (week 1 and 6 of intervention, and 3 months post intervention.)
  The CES-D scale is a well validated self-administered questionnaire used to measure depression. The 20 item scale has Likert scores ranging from "rarely or none of the time" (score 0), "some or little of the time" (score 1), "moderate or much of the time" (score 2), and "most or almost all the time" (score 3).Scores range from 0 to 60 with higher scores indicated greater depressive symptoms. A cut off at or above 20 has sensitivity 79% and specificity of 80% for major depression. Difference in CES-D measured at three time points (week 1 and 6 of the intervention and 3 months post intervention) will be reported and compared. The scale takes approximately 5-10 minutes to complete.
Differences in PROMIS-SD between time points | Three time points (week 1 and 6 of intervention, and 3 months post intervention.)
  The Participant Reported Outcomes Measurement Information System (PROMIS) Adult Short Form: Sleep Disturbance (PROMIS-SD), is an 8 item scale measuring overall sleep quality, disturbances, and satisfaction over the past 7 days on 5 point Likert scale with scores ranging from 1 to 5. Raw scores are converted into t scores ranging from 28.9 to 76.5, with higher scores indicating greater sleep disturbance. Exploratory analysis will compare scores at three time points (week 1 and 6 of the intervention and 3 months post intervention). The scale takes approximately 2 minutes to complete 26 and is available in Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Juarez-Reyes, MD, PhD, Study Director — Stanford University; Lisa Golman-Rosas, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zich JM, Attkisson CC, Greenfield TK. Screening for depression in primary care clinics: the CES-D and the BDI. Int J Psychiatry Med. 1990;20(3):259-77. doi: 10.2190/LYKR-7VHP-YJEM-MKM2. PMID 2265888
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Akman T, Yavuzsen T, Sevgen Z, Ellidokuz H, Yilmaz AU. Evaluation of sleep disorders in cancer patients based on Pittsburgh Sleep Quality Index. Eur J Cancer Care (Engl). 2015 Jul;24(4):553-9. doi: 10.1111/ecc.12296. Epub 2015 Mar 1. PMID 25727241
- [Background] Wu HS, Harden JK. Symptom burden and quality of life in survivorship: a review of the literature. Cancer Nurs. 2015 Jan-Feb;38(1):E29-54. doi: 10.1097/NCC.0000000000000135. PMID 24831042
- [Background] Chen D, Yin Z, Fang B. Measurements and status of sleep quality in patients with cancers. Support Care Cancer. 2018 Feb;26(2):405-414. doi: 10.1007/s00520-017-3927-x. Epub 2017 Oct 23. PMID 29058128
- [Background] Carlson LE. Mindfulness-based interventions for coping with cancer. Ann N Y Acad Sci. 2016 Jun;1373(1):5-12. doi: 10.1111/nyas.13029. Epub 2016 Mar 9. PMID 26963792
- [Background] Vollestad J, Nielsen MB, Nielsen GH. Mindfulness- and acceptance-based interventions for anxiety disorders: a systematic review and meta-analysis. Br J Clin Psychol. 2012 Sep;51(3):239-60. doi: 10.1111/j.2044-8260.2011.02024.x. Epub 2011 Sep 9. PMID 22803933
- [Background] Hoge EA, Bui E, Marques L, Metcalf CA, Morris LK, Robinaugh DJ, Worthington JJ, Pollack MH, Simon NM. Randomized controlled trial of mindfulness meditation for generalized anxiety disorder: effects on anxiety and stress reactivity. J Clin Psychiatry. 2013 Aug;74(8):786-92. doi: 10.4088/JCP.12m08083. PMID 23541163
- [Background] Schell LK, Monsef I, Wockel A, Skoetz N. Mindfulness-based stress reduction for women diagnosed with breast cancer. Cochrane Database Syst Rev. 2019 Mar 27;3(3):CD011518. doi: 10.1002/14651858.CD011518.pub2. PMID 30916356
- [Derived] Juarez-Reyes M, Martinez E, Xiao L, Goldman Rosas L. A Randomized Controlled Trial of a Culturally Adapted, Community-Based, Remotely Delivered Mindfulness Program for Latinx Patients With Breast Cancer is Acceptable and Feasible While Reducing Anxiety. Glob Adv Integr Med Health. 2024 Aug 16;13:27536130241274240. doi: 10.1177/27536130241274240. eCollection 2024 Jan-Dec. PMID 39157776